CLINICAL TRIAL: NCT02689713
Title: Prospective, Randomized, Double-blind Controlled Pilot Study to Compare Topical Voriconazole to Placebo as a Pain Reducing Agent at Skin Donor Sites
Brief Title: Pilot Study to Compare Topical Voriconazole to Placebo as a Pain Reducing Agent
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Inability to recruit subjects at the study site.
Sponsor: Kenneth Hargreaves (Other)
Collaborators: San Antonio Military Medical Center (U.S. Federal Agency); U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Kenneth Hargreaves, Chair, Dept. of Endodontics, The University of Texas Health Science Center at San Antonio
Organization: The University of Texas Health Science Center at San Antonio (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: HSC20120196H
Record Dates: First submitted 2016-02-04; First posted 2016-02-24 (Estimated); Last update posted 2018-12-17 (Actual); Status verified 2018-12

CONDITIONS: Pain; Thermal Injury; Burns; Hyperalgesia
Keywords: Burn Pain; Hyperalgesia; TRPV1; OLAMs
MeSH Terms: conditions — Pain; Burns; Hyperalgesia | interventions — Voriconazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Topical Voriconazole Study Drug Group (Experimental): Subjects between 18 and 60 years old who have sustained a burn wound of less than 30% total body surface area, or traumatic wounds requiring skin graft will have the Topical Voriconazole study drug placed on graft site.
  Interventions: Drug: Voriconazole (topical)
- Topical Sterile Water Placebo Group (Placebo Comparator): Subjects between 18 and 60 years old who have sustained a burn wound of less than 30% total body surface area, or traumatic wounds requiring skin graft will have the Topical Sterile Water Placebo placed on graft site.
  Interventions: Drug: Topical Sterile Water Placebo Group

INTERVENTIONS:
Drug: Voriconazole (topical) — The voriconazole (Vfend®-IV 200mg) will be applied topically to one of two skin graft sites at a concentration of 150 micromolar. Dialysates will be collected over 12 hours post-skin graft/voriconazole application for analysis in the lab of OLAM concentrations.
  Other Names: Vfend IV 200mg
  Arms: Topical Voriconazole Study Drug Group
Drug: Topical Sterile Water Placebo Group — Sterile water will be applied topically to the other of the two skin graft sites. Dialysates will be collected over 12 hours post-skin graft/sterile water application for analysis in the lab of OLAM concentrations.
  Other Names: Sterile Water Placebo
  Arms: Topical Sterile Water Placebo Group

SUMMARY:
This study seeks to test if the study drug (voriconazole), when applied topically to a burn wound on the skin will help to reduce pain.

DETAILED DESCRIPTION:
This single-center, prospective, randomized, double-blind, controlled pilot study conducted at San Antonio Military Medical Center will evaluate the effectiveness of topical voriconazole for pain relief at autogenous skin donor sites compared to a topical placebo application. The patients will act as their own control. All participants and investigators in the study will be blinded to the treatment arm utilized on each of the patient's donor sites (voriconazole versus placebo). Patients, who are scheduled for skin grafting and have met the inclusion criteria for this study, will be invited to enroll in the study. Only those patients who have been planned for skin graft sites that are approximately symmetrical in size will be allowed to enroll in the study. The donor site wounds will be studied using a paired design consisting of voriconazole or the placebo applied topically to same-patient matched donor sites. Patients will be queried via the pain assessment tool as to perceived pain at timed intervals. Dialysate samples will be collected via microdialysis probes at matching timed intervals in order to measure levels of oxidized linoleic acid metabolites shown in previous studies to be present in peripheral nerves.

ELIGIBILITY:
Inclusion Criteria:

1.1 Subject must be at least 18 years of age and no older than 60 years of age of either gender and in good general health.

1.2 Subject has sustained burn wounds of less than 30 percent of the total body surface area, in order to minimize the systemic effects on wound healing and the risk of infection (both of which increase with increasing burn size).

1.3 Subject has sustained Burn or trauma/orthopedic wounds do not involve the harvesting area.

1.4 Subject has sustained burn or trauma/orthopedic wounds that, in the judgment of the attending surgeon, require excision and grafting of sufficient extent to justify two donor sites of equal and symmetrical size on non-dependent body surfaces areas. Note: Only two donor sites will be studied, however if the subject requires more than two donor sites, they will not be excluded.

1.5 The scheduled excision and grafting procedure is the first such operation for the subject during this hospitalization and injury.

1.6 Subject agrees to participate in follow-up evaluations (Post Op Day 0-3 and one follow up appointment between Post Op day 30-45 for Donor site evaluation and photos of both donor sites.

Exclusion Criteria:

2.1 Critical illnesses such as those requiring ventilator support, or having a systemic infection or hemodynamic instability, defined as a mean arterial pressure less than 60 for an extended period of time or requiring vasoactive medications to support blood pressure.

2.2 Patients unable to accurately communicate pain secondary to medical illness, altered mental status, spinal cord injury, and known current narcotic drug use.

2.3 Patients unable to make his/her own decision for the informed consent. (Not seeking consent from the legal authorized representative; self consent only).

2.4 Major acute or chronic medical illnesses that could affect wound healing (e.g. peripheral vascular disease, blood clotting disorder).

2.6 Cellulitis or other infection of the potential donor sites.

2.7 Donor site has been previously harvested for grafting.

2.8 Donor site crosses a joint.

2.9 Any Corticosteroid use that could interfere with wound healing thus OLAM levels.

2.10 Subjects with greater than 30% total body surface area burns.

2.11 Pregnancy or lactation. (Beta HCG pregnancy test completed prior to operative procedure, not part of study) In the event that we have a record of a hysterectomy, no pregnancy test will be done, and the subject will be assumed NOT to be pregnant.

2.12 Prisoners.

2.13 Subjects having any contraindications for voriconazole. The contraindications are 1) known hypersensitivity to voriconazole; and 2) Coadministration of terfenadine, astemizole, cisapride, pimozide, quinidine or sirolimus, rifampin, carbamazepine, long acting barbiturates, high dose ritonavir, rifabutin, ergotamine, dihydroergotamine, oral contraceptives or St. John's Wort. A one week washout shall be determined for the above listed medications prior to allowing entry into the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2018-06-15 (Estimated); Primary Completion 2018-11-14 (Actual); Study Completion 2018-11-14 (Actual)

PRIMARY OUTCOMES:
Pain Levels reported by patient on the Four Point Category Pain Scale at specific timepoints over 72 hours will be compared to pre-operative baseline pain report. | Pre-operatively then over 72 hours post-skin graft procedure (1, 3, 6, 9, 12, 24, 36,48, 60 and 72 hours)
  Subjects will complete a pre-op pain assessment tool (Four Point Category Pain Scale consisting of 0-3 numeric with corresponding adjectives), then complete the same instrument at 1, 3, 6, 9, 12, 24, 36,48, 60 and 72 hours post-procedure.
Pain Levels reported by the patient on the Heft-Parker Pain Scale at specific timepoints over 72 hours will be compared to pre-operative baseline pain report. | Pre-operatively then over 72 hours post-skin graft (1, 3, 6, 9, 12, 24, 36,48, 60 and 72 hours)
  Subjects will complete a pre-op pain assessment tool (Heft-Parker Pain Scale - 170mm), then complete the same instrument at 1, 3, 6, 9, 12, 24, 36,48, 60 and 72 hours post-procedure.
Pain Levels reported by the patient on the Visual Analog Pain Scale at specific timepoints over 72 hours compared to pre-operative baseline pain report. | Pre-operatively then over 72 hours post-skin graft (1, 3, 6, 9, 12, 24, 36,48, 60 and 72 hours)
  Subjects will complete a pre-op pain assessment tool (Visual Analog Pain Scale - 100mm), then complete the same instrument at 1, 3, 6, 9, 12, 24, 36,48, 60 and 72 hours post-procedure.
Cutaneous dialysate levels collected over time to measure baseline vs. timepoint oxidized linoleic acid metabolites (OLAMs) levels. | Over 72 hours post-skin graft (1, 3, 6, 9, 12, 24, 36,48, 60 and 72 hours)
  Microdialysates will be collected from the CMA-70 probe and CMA-106 pump at 1, 2, 3, 6, 9,12, 24, 36, 48,60, and 72 hours post drug administration [+/- 20 minutes per time interval]. The specific timepoint dialysates levels will be analysed and compared to baseline.

SECONDARY OUTCOMES:
Skin graft donor site wounds compared for cosmetic healing via photograph at post-op visit | At scheduled post-op visit between 30-45 days post-procedure
  Digital photographs of the wounds will be taken at the post-op visit scheduled between 30-45 days after the skin graft procedure to assess the cosmetic appearance of the two wound sites.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher E White, MD, Principal Investigator — Brook Army Medical Center
Locations (1):
- San Antonio Military Medical Center, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share data.